CLINICAL TRIAL: NCT01127815
Title: Identify the Clinical Significance and Potential Implications of PWC in Patients With Pancreatic Cancer
Brief Title: Identify the Clinical Significance and Potential Implications of Peritoneal Washing Cytology (PWC) in Patients With Pancreatic Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Ching-Yao Yang, National Taiwan university Hospital
Other Study IDs: 201004002R
Record Dates: First submitted 2010-05-20; First posted 2010-05-21 (Estimated); Last update posted 2010-05-21 (Estimated); Status verified 2010-05

CONDITIONS: Pancreatic Cancer
Keywords: Peritoneal washing cytology; pancreatic cancer; peritoneal metastasis; anoikis; to determine the relationship between PWC results and clinicopathologic parameters of pancreatic cancers; to identify the predictive value of PWC and postoperative drainage cytology on the peritoneal recurrence or outcomes; to dissect the molecular mechanism of peritoneal recurrence, especially on the PWC-inducing peritoneal seeding process.
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control
Biospecimen Retention: Samples With DNA — peritoneal washing cells, postoperative drainage, and parts of tumor tissues
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Pancreatic cancer is a disease with an extremely poor prognosis. Such poor results are largely due to a high incidence of local or peritoneal recurrence even after curative R0 resection. If occult microscopic metastasis or residual cancer could be predicted correctly and identify the high risk of peritoneal recurrence, we may have chance to treat these patients by different multimodal locoregional or adjuvant therapy to improve the treatment outcome.

DETAILED DESCRIPTION:
The purpose of this study has three specific aims: (1) to determine the relationship between peritoneal washing cytology (PWC) results and clinicopathologic parameters of pancreatic cancers, (2) to identify the predictive value of PWC and postoperative drainage cytology on the peritoneal recurrence or outcomes, (3) to dissect the molecular mechanism of peritoneal recurrence, especially on the PWC-inducing peritoneal seeding process.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pancreatic cancers, other non-ductal pancreatic cancers , and benign pancreatic tumors (as negative control population) operated in Surgical Department after IRB proof and receiving patients' informed consent.

Exclusion Criteria:

* Pregnant women

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: operated in Surgical Department of National Taiwan University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2010-03; Primary Completion 2011-03 (Estimated); Study Completion 2011-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Yao Yang, M.D., Principal Investigator — National Taiwan University Hospital